CLINICAL TRIAL: NCT00907712
Title: Cardiovascular Assessment Before and After Limb Amputation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Department difficulties
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: orit semana, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-09
Record Dates: First submitted 2009-05-18; First posted 2009-05-22 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Diagnostic Techniques, Cardiovascular
Keywords: amputation; vascular; below knee; above knee; cardiovascular; echo; cardiovascular assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cardiovascular (No Intervention): cardiac echo
  Interventions: Other: cardiac echo examination

INTERVENTIONS:
Other: cardiac echo examination — cardiac echo examination - before and after the surgery

SUMMARY:
Vascular lower limb amputees have an increased morbidity and mortality. The aim of the study is to evaluate the hemodynamic changes after amputation and its relation to outcome.

ELIGIBILITY:
Inclusion Criteria:

* all vascular or diabetic patients before leg amputation

Exclusion Criteria:

* traumatic amputation
* sepsis patient
* urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
cardiovascular assessment | week

SECONDARY OUTCOMES:
complications | month

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

REFERENCES:
- [Background] Izumi Y, Satterfield K, Lee S, Harkless LB. Risk of reamputation in diabetic patients stratified by limb and level of amputation: a 10-year observation. Diabetes Care. 2006 Mar;29(3):566-70. doi: 10.2337/diacare.29.03.06.dc05-1992. PMID 16505507
- [Background] Izumi Y, Satterfield K, Lee S, Harkless LB, Lavery LA. Mortality of first-time amputees in diabetics: a 10-year observation. Diabetes Res Clin Pract. 2009 Jan;83(1):126-31. doi: 10.1016/j.diabres.2008.09.005. Epub 2008 Dec 20. PMID 19097667
- [Background] Remes L, Isoaho R, Vahlberg T, Hiekkanen H, Korhonen K, Viitanen M, Rautava P. Major lower extremity amputation in elderly patients with peripheral arterial disease: incidence and survival rates. Aging Clin Exp Res. 2008 Oct;20(5):385-93. doi: 10.1007/BF03325142. PMID 19039278
- [Background] Papazafiropoulou A, Tentolouris N, Soldatos RP, Liapis CD, Dounis E, Kostakis AG, Bastounis E, Katsilambros N. Mortality in diabetic and nondiabetic patients after amputations performed from 1996 to 2005 in a tertiary hospital population: a 3-year follow-up study. J Diabetes Complications. 2009 Jan-Feb;23(1):7-11. doi: 10.1016/j.jdiacomp.2007.11.008. Epub 2008 Apr 16. PMID 18413176